CLINICAL TRIAL: NCT01349855
Title: A Randomized, Double-blind, 2x2 Cross-over Euglycemic Clamp Study in Two Parallel Cohorts to Assess the Safety and Tolerability of Two Dose Levels of a New Formulation of Insulin Glargine and to Compare Its Pharmacodynamic and Pharmacokinetic Properties With 0.4 U/kg/Day Lantus® in an 8-days Multiple Dosing Regimen in Patients With Diabetes Mellitus Type 1
Brief Title: Repeated Dosing Study With a New Insulin Glargine Formulation and Lantus® in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TDR11626; 2010-023771-26 (EudraCT Number)
Record Dates: First submitted 2011-04-15; First posted 2011-05-09 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Dose Level 1
  Interventions: Drug: Insulin glargine HOE901
- Cohort 2 (Experimental): Dose Level 2
  Interventions: Drug: Insulin glargine HOE901

INTERVENTIONS:
Drug: Insulin glargine HOE901 — Pharmaceutical form:solution for injection: new formulation and marketed formulation Route of administration: subcutaneous

SUMMARY:
Primary Objective:

To assess the safety and tolerability of two dose levels of a new insulin glargine formulation in a once-daily multiple dosing regimen

Secondary Objective:

To compare the pharmacokinetic and pharmacodynamic properties of two dose levels of a new insulin glargine formulation with 0.4 U/kg Lantus® in a once-daily multiple dosing regimen

DETAILED DESCRIPTION:
The study duration per patient will be 33 to 68 days including 2 treatment periods of 10 days each separated by a wash-out period of 7-21 days.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects, between 18 and 65 years of age, inclusive, with diabetes mellitus type 1 for more than one year, as defined by the American Diabetes Association
* Body weight between 50.0 kg and 110.0 kg,
* Body Mass Index between 18.0 and 30.0 kg/m2 inclusive
* Stable insulin regimen for at least 2 months prior to study
* Certified as otherwise healthy for Type-1 Diabetes mellitus patient by assessment of medical history and physical examination
* Women of childbearing potential must have a negative pregnancy test and must use a highly effective method of birth control. During the entire study female subjects of child bearing potential must use two independent methods of contraception. The accepted double contraception methods include use of an intra-uterine device or hormonal contraception in addition to one of the following contraceptive options: 1) condom; 2) diaphragm; cervical/vault cap; 3) spermicide.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic (apart from diabetes mellitus type 1), hematological, neurological, psychiatric, systemic (affecting the body as a whole), ocular, gynecologic (if female), or infectious disease; any acute infectious disease or signs of acute illness
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months
* Presence or history of a drug allergy or clinically significant allergic disease according to the Investigator's judgment
* Participation in a trial with any investigational drug during the past three months
* Symptoms of a clinically significant illness in the 3 months before the study, which, according to the investigator's opinion, could interfere with the purposes of the study
* Regular use of any medication other than insulins in the last month before study start with the exception of thyroid hormones, lipid-lowering and antihypertensive drugs, and, if female, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days
* Known hypersensitivity to insulin glargine or excipients of the study drug
* Any history or presence of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in first degree relatives (parents, siblings or children)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety in terms of adverse and serious adverse events, vital signs, ECG, safety laboratory | up to day 10 of each period

SECONDARY OUTCOMES:
Glucose infusion rate | up to day 10 of each period
Pharmacokinetic parameter : Cmax | up to day 10 of each period
Pharmacokinetic parameter : Tmax | up to day 10 of each period
Pharmacokinetic parameter : AUC | up to day 10 of each period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site number 276001, Neuss, Germany

REFERENCES:
- [Derived] Becker RH, Dahmen R, Bergmann K, Lehmann A, Jax T, Heise T. New insulin glargine 300 Units . mL-1 provides a more even activity profile and prolonged glycemic control at steady state compared with insulin glargine 100 Units . mL-1. Diabetes Care. 2015 Apr;38(4):637-43. doi: 10.2337/dc14-0006. Epub 2014 Aug 22. PMID 25150159